CLINICAL TRIAL: NCT05638958
Title: Effect of Peri-implant Gap Grafting and Immediate Provisionalization With Customized Healing Abutments on the Stability of Peri-implant Soft Tissues - a Randomized Clinical Trial
Brief Title: Immediate Implants With Customized Abutments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Alexandre Perez, Dr, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AB0005
Record Dates: First submitted 2022-11-15; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Edentulous Alveolar Ridge Atrophy
Keywords: immediate implants; immediate provvisional; soft tissue recession

STUDY DESIGN:
Intervention Model Description: Test: A customized PEEK abutment mimicking the subgingival emergence of the extracted tooth will be screw retained on top of the implant to seal the extraction site.
  Control: A commercially available healing abutment will be screwed on top of the implant and a collagen sponge will be used to protect the graft.
Who Masked: Participant
Masking Description: The participants ant the biostatician will be blinded on the assignment group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): A customized PEEK abutment mimicking the subgingival emergence of the extraction site will be screw-retained on the implant to seal the extraction site and to support healing of buccal soft tissues.
  Interventions: Device: Immediate post-extractive Implant placement
- Control group (Active Comparator): A commercially available healing abutment will be screwed on top of the implant and a collagen sponge will be used to protect the graft.
  Interventions: Device: Immediate post-extractive Implant placement

INTERVENTIONS:
Device: Immediate post-extractive Implant placement — Teeth scheduled for extraction will be used to study the effect of a customized healing abutment. All patients should receive prophylactic antibiotic therapy of 2g of amoxicillin (or clindamycin 600mg if allergic to penicillin) 1 hour before the surgery. Implant placed along the lingual/palatal bone plate and the implant platform should be placed at the level of the buccal bone plate. GUIDOR easy-graft CRYSTAL will be used to fill the defect between implant and buccal bone plate, subsequently, a standard healing abutment or a customized healing abutment will be screw-retained on the implants.

SUMMARY:
Tooth extraction is followed by marked alterations of the tissue volume. The resorption process of at least the surrounding mucosa can be altered by using immediate implant placement and additional features such as immediate provisional crown, platform switching and grafting the gap between implant and buccal bone plate. The support of the gingival margin with a provisional crown led to an increase of buccal gingival tissue.

Teeth scheduled for extraction will be used to study the effect of a customized healing abutment.

The following groups will be randomly assigned:

Control: A commercially available healing abutment will be screwed on top of the implant and a collagen sponge will be used to protect the graft.

Test: A customized PEEK abutment mimicking the subgingival emergence of the extracted tooth will be screw retained on top of the implant to seal the extraction site.

DETAILED DESCRIPTION:
Tooth extraction is followed by marked alterations of the tissue volume. Incorporation of biomaterials into a fresh extraction socket can significantly reduce alveolar resorption but is not able to diminish the biologic process of the buccal bone plate. The resorption process of at least the surrounding mucosa can be altered by using immediate implant placement and additional features such as immediate provisional crown, platform switching and grafting the gap between implant and buccal bone plate. The support of the gingival margin with a provisional crown led to an increase of buccal gingival tissue. Platform switching seems to be a viable option to reduce interproximal bone level alterations and to limit the buccal soft tissue recession. Furthermore, augmenting the defect between the implant and the buccal bone plate has been proven to reduce the resorption process and lead to less shrinkage.

The primary objective is:

- The implant success

The Secondary objectives are:

* The Changes in mid-facial mucosal recession
* The changes in papilla height
* The changes in soft tissue ridge width
* The aesthetic evaluation
* The implant stability

ELIGIBILITY:
Inclusion Criteria:•

* The patient is ≥ 18 years old
* Extraction of single rooted tooth with healthy adjacent teeth (PD<5mm, no BOP)
* Patient must be able to understand the purpose of the study and to sign the consent form

Exclusion Criteria:

* Smoking status of more than 10 cigarettes/day
* History of uncontrolled metabolic disorders (e.g. diabetes mellitus)
* History of malignancy, radiotherapy, or chemotherapy
* Pregnant or breast feeding
* History of immunodeficiences
* existence of metabolic bone disease or disease affecting bone healing
* untreated or active periodontitis (BOP and PD>5mm)
* absence or defects of the buccal bone plate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2023-03-10 (Estimated)

PRIMARY OUTCOMES:
Implant success | 1 year of follow up
  Evaluated according to the criteria of Albrektsson et al. (1986):
  * the implant is immobile when tested clinically
  * Radiography does not demonstrate evidence of peri-implant radiolucency
  * Bone loss that is less than 0.2 mm annually after the implant's first year of service
  * No pain, discomfort or infection
Peri-implant marginal bone level- Radiographic Measurements | 1 year of follow up
  Peri-implant bone level will be assessed based on individual peri-apical x-rays performed at baseline, after implant placement, at the time of final impression at 90 days and after insertion of the definitive crown after 160 days using an individualized impression tray with resin imprints and at 1, 2, 3 years of follow up. The radiographic measurements will be performed by an independent evaluator, who will be unware of the assigned treatment.
Peri-implant marginal bone level- Radiographic Measurements | 2 years of follow up
  Peri-implant bone level will be assessed based on individual peri-apical x-rays performed at baseline, after implant placement, at the time of final impression at 90 days and after insertion of the definitive crown after 160 days using an individualized impression tray with resin imprints and at 1, 2, 3 years of follow up. The radiographic measurements will be performed by an independent evaluator, who will be unware of the assigned treatment.
Peri-implant marginal bone level- Radiographic Measurements | 3 years of follow up
  Peri-implant bone level will be assessed based on individual peri-apical x-rays performed at baseline, after implant placement, at the time of final impression at 90 days and after insertion of the definitive crown after 160 days using an individualized impression tray with resin imprints and at 1, 2, 3 years of follow up. The radiographic measurements will be performed by an independent evaluator, who will be unware of the assigned treatment.
Implant success | 2 years of follow up
  Evaluated according to the criteria of Albrektsson et al. (1986):
  * the implant is immobile when tested clinically
  * Radiography does not demonstrate evidence of peri-implant radiolucency
  * Bone loss that is less than 0.2 mm annually after the implant's first year of service
  * No pain, discomfort or infection
Implant success | 3 years of follow up
  Evaluated according to the criteria of Albrektsson et al. (1986):
  * the implant is immobile when tested clinically
  * Radiography does not demonstrate evidence of peri-implant radiolucency
  * Bone loss that is less than 0.2 mm annually after the implant's first year of service
  * No pain, discomfort or infection

SECONDARY OUTCOMES:
Changes in mid-facial mucosal recession | 1 year of follow up
  The height of the mid-facial mucosa will be measured using the drilling template at baseline before tooth extraction after implant placement at day 45±5 (wound healing day 160±5 (primary endpoint - impression for final restoration) and at 1, 2, 3 years of follow up. Changes of mid-facial mucosal recession will be drawn by subtracting the post-op measurements from the baseline measurements.
Changes in mid-facial mucosal recession | 2 years of follow up
  The height of the mid-facial mucosa will be measured using the drilling template at baseline before tooth extraction after implant placement at day 45±5 (wound healing day 160±5 (primary endpoint - impression for final restoration) and at 1, 2, 3 years of follow up. Changes of mid-facial mucosal recession will be drawn by subtracting the post-op measurements from the baseline measurements.
Changes in mid-facial mucosal recession | 3 years of follow up
  The height of the mid-facial mucosa will be measured using the drilling template at baseline before tooth extraction after implant placement at day 45±5 (wound healing day 160±5 (primary endpoint - impression for final restoration) and at 1, 2, 3 years of follow up. Changes of mid-facial mucosal recession will be drawn by subtracting the post-op measurements from the baseline measurements.
Changes in papilla height | 1 year of follow up
  Height of the mesial and distal papilla will be assessed by measuring the distance between the incisal edge and the tip of the papilla using a caliper to the nearest 0.5mm before tooth extraction, after implant placement 45±5 during wound healing and at the time of final impression at 90±5 days, at 160±14 days after insertion of the definitive crown and at 1, 2, 3 years of follow up. Papilla height changes will be assessed by subtracting post-op measurements from baseline measurements before tooth extraction or after implant placement.
Changes in papilla height | 2 years of follow up
  Height of the mesial and distal papilla will be assessed by measuring the distance between the incisal edge and the tip of the papilla using a caliper to the nearest 0.5mm before tooth extraction, after implant placement 45±5 during wound healing and at the time of final impression at 90±5 days, at 160±14 days after insertion of the definitive crown and at 1, 2, 3 years of follow up. Papilla height changes will be assessed by subtracting post-op measurements from baseline measurements before tooth extraction or after implant placement.
Changes in papilla height | 3 years of follow up
  Height of the mesial and distal papilla will be assessed by measuring the distance between the incisal edge and the tip of the papilla using a caliper to the nearest 0.5mm before tooth extraction, after implant placement 45±5 during wound healing and at the time of final impression at 90±5 days, at 160±14 days after insertion of the definitive crown and at 1, 2, 3 years of follow up. Papilla height changes will be assessed by subtracting post-op measurements from baseline measurements before tooth extraction or after implant placement.
Changes in soft tissue ridge width - Volumetric measurements | 1 year of follow up
  Digital scans of the implant region will be obtained at baseline before tooth extraction and after implant placement, at day 45±5 during wound healing of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Changes in soft tissue ridge width - Volumetric measurements | 2 years of follow up
  Digital scans of the implant region will be obtained at baseline before tooth extraction and after implant placement, at day 45±5 during wound healing of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Changes in soft tissue ridge width - Volumetric measurements | 3 years of follow up
  Digital scans of the implant region will be obtained at baseline before tooth extraction and after implant placement, at day 45±5 during wound healing of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Aesthetic evaluation (PES) | 1 year of follow up
  Pink esthetic score will be assessed on photographic images the tooth after final restoration and the insertion of the definitive crown. The assessment will be performed by an independent evaluator unaware of the assigned treatment.
Aesthetic evaluation (PES) | 2 years of follow up
  Pink esthetic score will be assessed on photographic images the tooth after final restoration and the insertion of the definitive crown. The assessment will be performed by an independent evaluator unaware of the assigned treatment.
Aesthetic evaluation (PES) | 3 years of follow up
  Pink esthetic score will be assessed on photographic images the tooth after final restoration and the insertion of the definitive crown. The assessment will be performed by an independent evaluator unaware of the assigned treatment.
Implant stability (ISQ) | 90 days after insertion of the definitive crown
  Implant stability will be assessed using a resonance frequency measurement device and assessing Implant Stability Quotient (ISQ) scores after implant placement, at the time of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Implant stability (ISQ) | 160 days after insertion of the definitive crown
  Implant stability will be assessed using a resonance frequency measurement device and assessing Implant Stability Quotient (ISQ) scores after implant placement, at the time of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Implant stability (ISQ) | 1 year of followup
  Implant stability will be assessed using a resonance frequency measurement device and assessing Implant Stability Quotient (ISQ) scores after implant placement, at the time of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Implant stability (ISQ) | 2 years of follow up
  Implant stability will be assessed using a resonance frequency measurement device and assessing Implant Stability Quotient (ISQ) scores after implant placement, at the time of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.
Implant stability (ISQ) | 3 years of follow up
  Implant stability will be assessed using a resonance frequency measurement device and assessing Implant Stability Quotient (ISQ) scores after implant placement, at the time of final impression at 90 days, at 160 days after insertion of the definitive crown and at 1, 2, 3 years of follow up.

CONTACTS AND LOCATIONS:
Locations (1):
- HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No